CLINICAL TRIAL: NCT00783406
Title: A Phase 2A, Double Blind (3rd Party Open), 4 Way Cross-Over, Placebo Controlled Study To Investigate The Pharmacokinetics, Safety, Toleration And Efficacy Of Single Inhaled Doses Of PF-00610355 In Moderate COPD Patients.
Brief Title: Safety, Toleration and Efficacy of Single Inhaled Doses of PF-00610355 in Chronic Obstructive Pulmonary (COPD) Patients.
Acronym: A7881010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A7881010
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — N-((4'-hydroxybiphenyl-3-yl)methyl)-2-(3-(2-((-2-hydroxy-2-(4-hydroxy-3-((methylsulfonyl)amino)phenyl)ethyl)amino)-2-methylpropyl)phenyl)acetamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF- 00610355 (Experimental)
  Interventions: Drug: PF-00610355
- PF-00610355 (Experimental)
  Interventions: Drug: PF-00610355
- PF -00610355 (Experimental)
  Interventions: Drug: PF-00610355
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00610355 — dry powder inhaler, 1472 mcg, single dose
  Arms: PF- 00610355
Drug: PF-00610355 — dry powder inhaler, 736 mcg, single dose
  Arms: PF-00610355
Drug: PF-00610355 — dry powder inhaler, 368 mcg, single dose
  Arms: PF -00610355
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will look at the pharmacokinetics, safety, toleration and efficacy of PF-00610355 in the chronic obstructive pulmonary disease (COPD) population. The doses in this study are intended to explore the anticipated clinical dose range.

ELIGIBILITY:
Inclusion Criteria:

* Post-bronchodilator FEV1/ FVC ratio of <0.7.
* Post bronchodilator FEV1 of 50-80% (inclusive) of predicted.
* Body Mass Index (BMI) of less than 35 kg/m2; and a total body weight greater that 40 kg.
* Current smokers, or ex-smokers who have abstained from smoking for at least 6 months.

Exclusion Criteria:

* Subjects having more than 2 exacerbations requiring treatment with oral steroids or hospitalization for the treatment of COPD in the previous year.
* History of lower respiratory tract infection or significant disease instability during the month preceding screening or during the period between screening and randomization.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To characterize the single dose pharmacokinetics of inhaled PF-00610355 in COPD patients. | up to 8 days post dose
To evaluate the safety & toleration of single inhaled doses of PF-00610355 in COPD patients | up to 24 hours post dose

SECONDARY OUTCOMES:
To investigate the efficacy of a single inhaled dose of PF-00610355 in COPD patients. | up to 24 hours post dose
To investigate the exposure/response relationship of PF-00610355. | up to 8 days post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Wiesbaden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7881010&StudyName=Safety%2C%20Toleration%20and%20Efficacy%20of%20Single%20Inhaled%20Doses%20of%20PF-00610355%20in%20Chronic%20Obstructive%20Pulmonary%20%28COPD%29%20Patients.